CLINICAL TRIAL: NCT07223060
Title: A Randomized, Single-center, Two-cell, Double-blind and Parallel-group Design Clinical Study Conducted in the Bangkok, Thailand Area, to Investigate the Clinical Efficacy of a Test Toothpaste Containing 0.454% Stannous Fluoride as Compared to a Regular Fluoride Toothpaste Containing 0.76% Sodium Monofluorophosphate in Controlling Supragingival Calculus Formation Over a 12-week Period.
Brief Title: Efficacy of Toothpaste Containing 0.454% Stannous Fluoride as Compared to a Regular Fluoride Toothpaste Containing 0.76% Sodium Monofluorophosphate in Controlling Supragingival Calculus Formation Over a 12-week Period.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2017-04-TAR-SNDZ-YPZ
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Calculus, Dental
MeSH Terms: conditions — Dental Calculus | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test 1 toothpaste (Experimental)
  Interventions: Drug: 0.454% stannous fluoride
- Test 2 toothpaste (Active Comparator)
  Interventions: Drug: 0.76% sodium monofluorophosphate

INTERVENTIONS:
Drug: 0.454% stannous fluoride — brushed twice daily, morning and evening for 2 minutes eact time
  Arms: Test 1 toothpaste
Drug: 0.76% sodium monofluorophosphate — brushed twice daily, morning and evening for 2 minutes eact time
  Arms: Test 2 toothpaste

SUMMARY:
To evaluate the comparative clinical efficacy of a test toothpaste containing 0.454% stannous fluoride as compared to a regular fluoride toothpaste containing 0.76% sodium monofluorophosphate in controlling supragingival calculus formation over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were required to sign an Informed Consent form
* Subjects had to be in general good health
* Male and female adults between the ages of 18-70 (inclusive)
* Six (6) scoreable mandibular anterior teeth free of large restorations or dental prosthetic crowns
* Subjects were required to possess a Volpe-Manhold Calculus Index of at least 7.0
* Subjects had to be able to participate for the full duration (20 weeks) of the study

Exclusion Criteria:

* Presence of orthodontic appliances or removable prosthesis at the lower jaw or more than one mandibular anterior tooth with a prosthetic crown or veneer
* Tumor(s) or significant pathology of the soft or hard tissues of the oral cavity
* Moderate or advanced periodontal disease
* Five or more carious lesions requiring immediate care
* Use of antibiotics or steroids any time during one month prior to entry into the study
* Participation in any other clinical study or panel test
* Pregnant or breast feeding women
* History of allergies to dentifrice and personal care ingredients
* Allergies to dentifrice products
* Medical reasons that prohibit eating or drinking for 4 hours prior to clinical facility visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Supragingival calculus formation via Volpe-Manhold Calculus Index | baseline and 12 week measurement
  index for comparing the amount of dental calculus

CONTACTS AND LOCATIONS:
Overall Officials: Dutmanee Seriwatanachai, Principal Investigator — Mahidol University
Locations (1):
- M U International Oral Science Research, Ltd., Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No